CLINICAL TRIAL: NCT05434897
Title: A Randomized, Double-blind, Placebo Self-controlled Phase I/II Clinical Study to Evaluate the Safety, Tolerability and Preventive Efficacy of AK3280 Cream After Cicatrectomy in Patients With Hypertrophic Scar in China.
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of AK3280 Cream on Hypertrophic Scar
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK3287-2001
Record Dates: First submitted 2022-06-16; First posted 2022-06-28 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2% dose AK3280 cream (Experimental): After the 4-week screening period, Eligible subjects will be administered daily 2% dose AK3280 cream b.i.d. for 12weeks.
  Interventions: Drug: AK3280 Cream
- 4% dose AK3280 cream (Experimental): After the 4-week screening period, Eligible subjects will be administered daily 4% dose AK3280 cream b.i.d. for 12weeks.
  Interventions: Drug: AK3280 Cream
- 8% dose AK3280 cream (Experimental): After the 4-week screening period, Eligible subjects will be administered daily 8% dose AK3280 cream b.i.d. for 12weeks.
  Interventions: Drug: AK3280 Cream
- Placebo cream (Active Comparator): The same subject will be randomized to receive topical administration of AK3280 cream or placebo cream at S1 and S3, respectively.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: AK3280 Cream — Active Substance: AK3280, Pharmaceutical Form:Cream, Route of Administration: External use
  Other Names: AK3287
  Arms: 2% dose AK3280 cream; 4% dose AK3280 cream; 8% dose AK3280 cream
Drug: Placebo cream — Active Substance: Placebo, Pharmaceutical Form: Cream, Route of Administration: External use
  Arms: Placebo cream

SUMMARY:
A randomized, double-blind, placebo self-controlled phase I/II clinical study to evaluate the safety, tolerability and preventive efficacy of different doses of AK3280 cream （AK3287 ） after cicatrectomy in Patients with Hypertrophic Scar in China.

DETAILED DESCRIPTION:
Thirty patients with hypertrophic scar who will scheduled for cicatrectomy and meet the all inclusion criteria and none of exclusion criteria will participate in this study. There will be 3 cohorts for 2%, 4%, 8% doses of AK3287 （AK3280 cream） in turn, and 10 participants in each cohort. Participants in every cohort will receive cicatrectomy on day -5, and their incisions will be divided into 3 parts with equal length after length measurement on day 1, named S1, S2, S3. S1 is proximal, and S3 is distal. AK3280 cream （AK3287 ） or placebo will topically administrated to S1 or S3 randomly, twice a day (BID). In this study, S1 and S3 paired, placebo self-control design will be adopted.

The study includes a 4-week screening period, a 12-week drug observation period, and a 2-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients who sign informed consent before participating in the study.
* 2) Patients aged between 18 and 60 (including 18 and 60).
* 3)Patients who understand and be willing to follow the study procedure and be able to complete the whole process of the study.
* 4) Patients with visible hypertrophic scars in any location other than the face and anterior middle and upper neck caused by trauma or surgery and planned for surgical treatment.
* 5) Patients with postoperative scar length ≥ 6 cm, and preoperative scar length ≥4cm.
* 6) Women of childbearing age should have negative serum pregnancy test during screening period and on study day 1.

Exclusion Criteria:

* 1) Patients who were systematically treated or topically treated with corticosteroids or immunosuppressants during the 30 days prior to the screening period;
* 2) Patients who accepted systematically chemotherapy during 30 days prior to the screening period;
* 3) Patients whose hypertrophic scars are being locally infected, or with sepsis;
* 4) Hypertrophic scar patients with potential keloid trend or keloid history;
* 5) Patients with autoimmune diseases or immune insufficiency or defects
* 6)Patient with uncontrolled diabetes - HbA1c (glycosylated hemoglobin A1c) ≥ 8% ，with peripheral neuropathy, peripheral arterial atresia, or other vascular diseases;
* 7) Patients with abnormal anticoagulation or coagulation function;
* 8) Patients with atrophic skin diseases, rheumatism or hemopathy ;
* 9) Patients with abnormal liver and kidney function: I. AST (Aspartate Transaminase) or ALT (Alanine Transaminase) > the upper limit of normal, and total bilirubin > the upper limit of normal; Ii. AST or ALT≥1.5 times of the upper limit of normal; Iii. Creatinine clearance rate< 60mL/ min ;
* 10) Patients with infectious diseases such as positive antibody of HBV (hepatitis B virus) , HCV (hepatitis B virus), HIV (human immunodeficiency virus) or syphilis;
* 11) The patients or their family have a history of hypersensitivity or allergies to multiple substances, or serious atopic dermatitis, or are not suitable for participate this study by investigator's judgment;
* 12) Patients who are currently or possibly suffering from malignant tumors;
* 13) Patients with definite diagnosis of mental illness with irregular medication;
* 14) Patients received any treatment that may affect wound healing, cicatrization, hemostasis or anti-coagulation, possible interactions with investigational drug within 30 days prior to randomization;
* 15) The investigators judge that patients have safety risk, or cannot complete this study or collect all blood concentration because of patient's general condition, comorbidity or medical history, or abnormal physical examination/vital signs/laboratory tests/electrocardiogram;
* 16) Patients who have received scar ablation or X-ray therapy within the past 6 months;
* 17) Patients have participated in other clinical trials of medicine or devices within 30 days prior to the screening period;
* 18) Pregnant or lactating women;
* 19) Women and men of reproductive age who are not willing to use highly effective contraception during the study period and at least 3 months after the last administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Assessment of adverse events（AE）/ serious adverse events (SAEs) | Up to 14 weeks
  Adverse Events occurring from day1 to last visit will be assessed and graded according to Common Terminology Criteria for Adverse Events version 5.0.
Number of participants with abnormal Skin Examination | Up to 14 weeks
  The skin examination should be performed under sufficient light and at room temperature , including skin lesion, inflammation, allergy, Scar hyperplasia.
Number of participants with abnormal vital signs | Up to 14 weeks
  Vital signs: include pulse, respiration, body temperature and blood pressure
Number of participants with abnormal Physical examination findings | Up to 14 weeks
  Physical examination ： include height, weight, head and neck, mouth, chest, abdomen, lymph nodes, nerves and mind, limbs and other sites
Number of participants with abnormal 12-lead ECG readings | Up to 14 weeks
Number of participants with abnormal laboratory test results | Up to 14 weeks
  Laboratory tests：include blood routine examination， blood biochemistry ，urine routine test and coagulation function

SECONDARY OUTCOMES:
Within 12 weeks of topical administration, the proportion of scar hyperplasia/recurrence compared in S1 and S3 segment | 4 weeks， 8 weeks, 12 weeks, and unscheduled visits (up to 14 weeks)
  There are 4 items in the VSS scale（Vancouver Scar Scale） , Vascularity、 Pigmentation、 Pliability and Height. A total of 13 points, with minimum 0 indicating normal skin and maximum 13 indicating the most scarring and worst appearance. Two trained and skilled physicians are required to objectively evaluate the scar of all subjects. The scar was observed after pressing with a special glass slide for 2 seconds, and the average score of both was used as the final score of VSS to reduce subjective bias.
  Scar hyperplasia/recurrence was defined as the Height item score of the VSS scale ≥2.
  If two investigators had different scores in Height item, for safety, the higher score would be final result.
Within 12 weeks of topical administration, the change of VSS （Vancouver Scar Scale ） total score compared in S1 and S3 segment from baseline | 4 weeks， 8 weeks, 12 weeks, and unscheduled visits (up to 14 weeks)
  There are 4 items in the VSS scale（Vancouver Scar Scale） , Vascularity、 Pigmentation、 Pliability and Height. A total of 13 points, with minimum 0 indicating normal skin and maximum 13 indicating the most scarring and worst appearance. Two trained and skilled physicians are required to objectively evaluate the scar of all subjects. The scar was observed after pressing with a special glass slide for 2 seconds, and the average score of both was used as the final score of VSS to reduce subjective bias.
Within 12 weeks of topical administration, the change of mean thickness by 3D photography compared in S1 and S3 segment from baseline | 4 weeks， 8 weeks, 12 weeks, and unscheduled visits (up to 14 weeks)
  Taking 5 points in each segment can automatically get the thickness of each point by 3D photography and calculate the average thickness.
Within 12 weeks of topical administration, the change of surface area per centimeter by 3D photography compared in S1 and S3 segment from baseline | 4 weeks， 8 weeks, 12 weeks, and unscheduled visits (up to 14 weeks)
  Surface area can be obtained directly by 3D photography，then calculate the surface area per centimeter.
Within 12 weeks of topical administration, the change of volume per centimeter by 3D photography compared in S1 and S3 segment from baseline | 4 weeks， 8 weeks, 12 weeks, and unscheduled visits (up to 14 weeks)
  Volume can be obtained directly by 3D photography，then calculate the volume per centimeter.
Within 12 weeks of topical administration, the change of blood flow in laser speckle imaging system compared in S1 and S3 segment from baseline | 4 weeks， 8 weeks, 12 weeks, and unscheduled visits (up to 14 weeks)
  Blood perfusion of capillary of scar, para-scar and normal tissue will be tested by laser speckle imaging system to evaluate scar recurrence compared S1 with S3.
Cmax (Maximum observed concentration) of AK3280 after topical administration of AK3280 onitment. | Up to 14 weeks
Ctrough (trough level concentration) of AK3280 after topical administration of AK3280 onitment. | Up to 14 weeks
Tmax (Time of peak plasma concentration) of AK3280 after topical administration of AK3280 onitment. | Up to 14 weeks
AUC0-t (Area under the concentration-time curve from time zero to the last measurable concentration ) of AK3280 after topical administration of AK3280 onitment. | Up to 14 weeks
CL/F (apparent clearance) of AK3280 after topical administration of AK3280 onitment. | Up to 14 weeks
Cmax of AK3280 M2 after topical administration of AK3280 onitment. | Up to 14 weeks
  Four metabolites (M1-M4) were detected in human plasma collected after oral administration of AK3280. M2 is the most abundant metabolite circulating in the blood, also found in urine.
Ctrough of AK3280 M2 after topical administration of AK3280 onitment. | Up to 14 weeks
Tmax of AK3280 M2 after topical administration of AK3280 onitment. | Up to 14 weeks
AUC0-t of AK3280 M2 after topical administration of AK3280 onitment. | Up to 14 weeks
CL/F of AK3280 M2 after topical administration of AK3280 onitment. | Up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jihong Liu, Study Director — Medical Director; Yan Wu, Study Chair — Chief Medical Officer
Locations (1):
- Shanghai Ninth People's Hospital,Shanghal JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No